CLINICAL TRIAL: NCT03265652
Title: Intense Pulsed Light and Meibomian Gland Expression (MGX) Versus MGX Alone in the Treatment of Dry Eye Disease Secondary to Meibomian Gland Dysfunction
Brief Title: IPL and MGX Versus MGX Alone in the Treatment of Dry Eye Disease Secondary to MGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUM-VBU-IPL-M22-17-02; 0171-17-SZMC (Other: Shaarei Zedek Hospital)
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction
Keywords: Intense Pulsed Light; Meibomian Gland Dysfunction; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to a study arm and a control arm. Subjects in the study arm will be treated with IPL and meibomian gland expression. Subjects in the control arm will be treated with sham and meibomian gland expression.
Who Masked: Participant
Masking Description: Subjects in the study arm will receive a series of IPL pulses using the M22 IPL handpiece. In subjects of the control arm, the device will be disabled. The subject will feel the lightguide on the skin, will hear clicking sounds, but no light will be actually produced by the M22 device. Since during treatment both eyes of the subject will be fully occluded, no subject will be able to see if the treatment is actual or sham. There is no way to completely mask the subjects, since the IPL generally causes slight redness of the skin, and in some patients is may also cause some discomfort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intense Pulsed Light (IPL) therapy (Experimental): Subjects with receive 10-15 intense pulsed light (IPL) pulses on the skin of the malar region (both cheeks, from tragus to tragus including the nose) and up to 3 mm from the lid margin of the lower eyelid. Following the administration of IPL pulses, subjects will undergo meibomian gland expression.
  Interventions: Device: Intense Pulsed Light (IPL) therapy
- Sham therapy (Placebo Comparator): Participants will undergo a sham treatment that will mimic the intense pulsed light (IPL) therapy. The tip of the IPL lightguide will be placed in 10-15 locations on the skin of the malar region (both cheeks, from tragus to tragus including the nose) and up to 3 mm from the lid margin of the lower eyelid, but IPL pulses will not be actually delivered. Following this sham procedure, subjects will undergo meibomian gland expression.
  Interventions: Device: Sham therapy

INTERVENTIONS:
Device: Intense Pulsed Light (IPL) therapy — Intense pulsed light therapy is a non-invasive and non-laser light treatment that is FDA-approved for various conditions in dermatology. Subjects will receive a total of 4 treatments over the course of the study, at intervals of 2 weeks. Each treatment will include applications on 10-15 IPL pulses in the malar region and close to the lower eyelids, followed by meibomian gland expression. Meibomian gland expression will be implemented by squeezing the meibomian glands with the aid of two Q-tips positioned on either side of the meibomian glands, or with a meibomian gland expressor forceps.
  Arms: Intense Pulsed Light (IPL) therapy
Device: Sham therapy — Subjects will receive a total of 4 treatments over the course of the study, at intervals of 2 weeks. Each treatment will include a sham application of IPL on 10-15 locations in the malar region and close to the lower eyelids, followed by meibomian gland expression. Meibomian gland expression will be implemented by squeezing the meibomian glands with the aid of two Q-tips positioned on either side of the meibomian glands, or with a meibomian gland expressor forceps.
  Arms: Sham therapy

SUMMARY:
The aim of the current study is to examine the contribution of intense pulsed light (IPL) for relieving signs and symptoms of dry eye due to meibomian gland dysfunction. The effect of IPL will be examined in a study designed as a randomized controlled trial. In the study arm, subjects will undergo 4 treatment sessions, consisting of IPL pulses immediately followed by expression of the meibomian glands. In the control arm, subjects will undergo the same treatments, except that the IPL pulses will be disabled. For each subject, the duration of the study will be 10 weeks, as explained in the detailed description,

DETAILED DESCRIPTION:
Outcome measures (tear break-up time, tear film osmolarity, meibomian gland assessment, number of meibomian glands yielding liquid secretion in lower eyelid , meibography, self-assessed symptoms and close up photos of the lid margins) will be measured at baseline. All subjects will receive 4 treatments at 2 weeks intervals. In each treatment session, a subject allocated to the study group will be treated with IPL administered in the malar region, from tragus to tragus including the nose, 2-3 mm below the lower eyelids. Immediately following the IPL administration, the meibomian glands will be manually expressed from both eyelids. Subjects in the control arm will receive exactly the same treatment, except that the IPL administration will be sham. A single follow-up will occur at 10 weeks after the baseline (or 4 weeks after the 4th treatment session). At the follow-up, the changes in the outcome measures will be evaluated, and compared between the two arms.

For each subject, the duration of the study will be 10 weeks: 1st treatment at baseline; 2nd treatment at 2 weeks after baseline; 3rd treatment at 4 weeks after baseline; 4th treatment at 6 weeks after baseline; and a single follow-up at 10 weeks after baseline).

Statistically significant differences between the two arms will support the study hypothesis that IPL treatment itself provides relief to both signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to read, understand and sign an Informed Consent (IC) form
2. Subject is 18 years or older
3. Subject has Fitzpatrick skin type I to IV
4. SPEED questionnaire equal or more than 10
5. OSDI questionnaire equal or more than 23
6. In both eyes, at least 5 non-atrophied meibomian glands on the lower eyelid.
7. In both eyes, Tear break up time equal or less than 7 seconds
8. In both eyes, MGA (the total meibomian gland score for 15 glands of the lower eyelid) is smaller or equal to 12

Exclusion Criteria:

1. Contact lens wear within the month prior to screening
2. Unwilling to discontinue use of contact lenses for the duration of the study
3. Ocular surgery or eyelid surgery within 6 months prior to screening
4. Neuro-paralysis in the planned treatment area within 6 months prior to screening
5. Other uncontrolled eye disorders affecting the ocular surface, for example active allergies
6. Current use of punctal plugs
7. Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
8. Uncontrolled infections or uncontrolled immunosuppressive diseases
9. Subjects with ocular infections within 6 months prior to screening
10. Prior history of cold sores or rashes in the perioral area or in the planned treatment area that could be stimulated by light at a wavelength of 560 nm to 1200 nm (e.g., Herpes simplex 1 & 2, Systemic Lupus erythematosus, porphyria)
11. Use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, such as Isotretinoin, Tetracycline, Doxycycline, or St. John's Wort within 3 months prior to screening
12. Over exposure to sun within 4 weeks prior to screening, in the judgment of the investigator
13. Administration of prescription eye drops for dry eye within 7 days prior to screening, excluding artificial tears and glaucoma drops
14. Radiation therapy to the head or neck within 12 months prior to screening, or planned radiation therapy within 8 weeks after completion of all IPL treatments
15. Treatment with chemotherapeutic agent within 8 weeks prior to screening, or planned chemotherapy within 8 weeks after completion of all IPL treatments
16. New topical treatments within the area to be treated, or oral therapies within 3 months prior to screening, except over-the-counter acetaminophen-based analgesics (such as Extra Strength Tylenol®) for pain management after study treatment, new oral omega 3 fatty acid supplements and topical artificial tears
17. Change in dosage of any systemic medication within 3 months prior to screening
18. Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up over the study period
19. Legally blind in either or both eyes
20. History of migraines, seizures or epilepsy
21. IPL treatment within 12 months prior to screening
22. Lipiflow treatment, or any other thermal treatment of the eyelids, within 6 months prior to screening
23. Expression of the meibomian glands within 6 months prior to screening
24. Any condition revealed during the eligibility screening process whereby the investigator deems the subject inappropriate for this study
25. Women below the age of menopause (50 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Change of baseline TBUT | 10 weeks
  Change of Tear break up time in the study eye, from baseline to follow-up

SECONDARY OUTCOMES:
Change from baseline MGA | 10 weeks
  Change of Meibomian gland secretion score, from baseline to follow-up, in both eyes
Change from baseline OSDI | 10 weeks
  Change of self-assessed symptoms with the OSDI questionnaire, from baseline to follow-up, in both eyes

OTHER OUTCOMES:
Change from baseline MGYLS | 10 weeks
  Change of the number of meibomian glands yielding liquid secretion, from baseline to the follow-up
Change from baseline TFO | 10 weeks
  Change of the tear film osmolarity, from baseline to the follow-up
Change from baseline Meiboscore | 10 weeks
  Change of the Meiboscore evaluated with meibography, from baseline to the follow-up
Percentage of study eyes with normal TBUT | 10 weeks
  Percentage of study eyes with TBUT > 10 seconds at the follow-up
Percentage of subjects with normal OSDI | 10 weeks
  Percentage of subjects with OSDI < 23 at the follow-up
Percentage of subjects with normal MGA | 10 weeks
  Percentage of eyes with MGA > 12 at the follow-up
Qualitative assessment of eyelid appearance | 10 weeks
  High resolution photos of the upper and lower eyelids in both eyes

CONTACTS AND LOCATIONS:
Overall Officials: David Zadok, MD, Principal Investigator — Shaarei Zedek Hospital ( Jerusalem)
Locations (1):
- Shaare Zedek, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
At this point it is not yet decided if and how to share IPD with other researchers